CLINICAL TRIAL: NCT05037942
Title: The Influence of Restriction Pressure on Indices of Exercise-Induced Muscle Damage Following Low-Load Blood Flow-Restricted Resistance Exercise: A Randomised Controlled Trial in Healthy Adults
Brief Title: The Effects of Restriction Pressure on Muscle Damage Responses to Blood Flow Restriction Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Surrey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: FHMS 20-21 151 EGA
Record Dates: First submitted 2021-08-31; First posted 2021-09-08 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Muscle Damage; Muscle Soreness; Muscle Strength
Keywords: Muscle Damage; Muscle Soreness; Muscle Strength; Blood Flow Restriction
MeSH Terms: conditions — Myalgia

STUDY DESIGN:
Intervention Model Description: The study uses a within-between, unilateral design, in which participants will be randomly allocated into one of two experimental groups using a stratified random allocation technique. Each group will perform blood flow-restricted exercise with one leg and the same exercise protocol without BFR with the contralateral leg. Experimental groups will be differentiated by the tourniquet pressure used during the BFR condition: i) tourniquet pressure set to 40% of limb occlusion pressure or ii) tourniquet pressure set to 80% of limb occlusion pressure. Legs will be counterbalanced such that the BFR and control conditions in each study group contain an equal number of dominant and non-dominant legs. This study design allows comparison between the two experimental conditions (i.e., 40% vs. 80% limb occlusion pressure), while allowing participants to serve as their own control condition.
Who Masked: Outcomes Assessor
Masking Description: Given the perceptual response that occurs under different occlusion pressures, it is difficult to mask the participant to the experimental conditions. Efforts will be made to minimise detection bias by blinding the outcome assessor to the study conditions and the timepoints from which the data has been collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Blood flow-restricted exercise at 40% limb occlusion pressure (BFR-40) (Experimental): Participants in BFR-40 will perform a lower-body exercise protocol under BFR set to 40% of the participants' relative limb occlusion pressure.
  Interventions: Other: Blood flow restriction at 40% limb occlusion pressure
- Blood flow-restricted exercise at 80% limb occlusion pressure (BFR-80) (Experimental): Participants in BFR-80 will perform the same lower-body BFR exercise protocol as BFR-40; however, the occlusion pressure will be set to 80% of the participants' relative limb occlusion pressure.
  Interventions: Other: Blood flow restriction at 80% limb occlusion pressure
- Control for BFR-40 (No Intervention): Participants randomised to BFR-40 will perform the same exercise protocol without BFR with the contralateral leg.
- Control for BFR-80 (No Intervention): Participants randomised to BFR-80 will perform the same exercise protocol without BFR with the contralateral leg.

INTERVENTIONS:
Other: Blood flow restriction at 40% limb occlusion pressure — A 13-cm-wide pneumatic cuff will be applied to the most proximal portion of the chosen thigh (as determined by randomisation), immediately distal to the inguinal fold, prior to a bout of lower-body resistance exercise. The cuff will be inflated to 40% of limb occlusion pressure pressure and will remain inflated throughout the exercise (total occlusion time: ~5 mins).
  Other Names: Vascular restriction; Vascular occlusion; Venous restriction
  Arms: Blood flow-restricted exercise at 40% limb occlusion pressure (BFR-40)
Other: Blood flow restriction at 80% limb occlusion pressure — A 13-cm-wide pneumatic cuff will be applied to the most proximal portion of the chosen thigh (as determined by randomisation), immediately distal to the inguinal fold, prior to a bout of lower-body resistance exercise. The cuff will be inflated to 80% of limb occlusion pressure pressure and will remain inflated throughout the exercise (total occlusion time: ~5 mins).
  Other Names: Vascular restriction; Vascular occlusion; Venous restriction
  Arms: Blood flow-restricted exercise at 80% limb occlusion pressure (BFR-80)

SUMMARY:
Blood flow restriction (BFR) exercise involves the application of a constriction device to the limbs to restrict muscle blood flow during exercise. In recent years, BFR has become increasingly popular due to its additive effects on low-load resistance training, often promoting greater increases in muscle strength and size compared to similar resistance training without BFR. However, like other exercise, it is possible that BFR exercise can cause exercise-induced muscle damage (EIMD) that results in short-term reductions in muscle function and increased muscle soreness and swelling. One major variable that may influence the onset of EIMD is the restriction pressure used to restrict blood flow; however, the influence of restriction pressure on resistance EIMD is unclear.

The purpose of this study is to investigate effects of two different restriction pressures (low and high) on EIMD responses to a bout of low-load BFR resistance exercise in a sample of healthy, active adults. It is hypothesised that a higher restriction pressure will result in increased EIMD compared to a lower restriction pressure. To test this hypothesis, participants will perform a lower-body exercise protocol with and without BFR, and several markers of EIMD will be assessed before and immediately, 24, 48, and 72 hours after the exercise.

DETAILED DESCRIPTION:
Following screening for the inclusion and exclusion criteria of the study, eligible participants will be fully informed of the study purposes and procedures and written consent will be acquired. During this study, participants will be randomly allocated into one of two experimental groups, with each group performing blood flow-restricted knee extension exercise with one leg and the same exercise protocol without BFR with the contralateral leg. Experimental groups will be differentiated by the tourniquet pressure used during the BFR condition. Several indirect markers of EIMD will be assessed at baseline and 24, 48, and 72 hours after the exercise bout. Additional neuromuscular assessments will be performed immediately post-exercise to provide insight into the fatiguability of the exercise protocol.

Participants will be required to attend the laboratory on five separate occasions: one visit for screening, assessment of limb occlusion pressure (i.e., the lowest pressure required to occlude blood flow to the limb), and familiarisation of the exercise protocol and neuromuscular assessments, one visit for completion of the exercise protocol and baseline/post-exercise tests, and three follow-up visits. All participants will be asked to refrain from alcohol and exercise from 24 hours prior to the exercise trial up to their final visit. The consumption of any pain-relieving medications (e.g., anti-inflammatory drugs) and undergoing of any muscle damage treatments (e.g., massage) will be prohibited throughout the study. To minimise the effects of pre-exercise feeding on the outcome measures, visits will be scheduled for the morning and participants will attend the lab following an overnight fast of a minimum of 10 hours, although water may be consumed ad libitum. All post-exercise measures will be collected at the same time of day ± 1 hours.

ELIGIBILITY:
Inclusion Criteria:

* Recreationally active (defined as performing ≥ 150 minutes of moderate-intensity or ≥ 75 minutes of vigorous-intensity exercise per week for the past 6 months)
* Resistance-untrained (defined as performing less than 2 resistance exercise sessions per week for the past 6 months)

Exclusion Criteria:

* Any history of cardiovascular (including hypertension [diastolic > 90 and/or systolic blood pressure > 140 mmHg] and peripheral arterial vascular disease), metabolic, respiratory (including severe asthma), haematological (including deep vein thrombosis and pulmonary embolism), neurological, gastrointestinal, kidney, liver, or musculoskeletal disease
* Current or previous musculoskeletal injury that may be aggravated by exercise
* Current smoker
* Recently used prescribed anti-inflammatory medication within the previous 1 month
* Self-reported or diagnosed menstrual irregularities within ≥ 3 months prior to recruitment
* Currently pregnant

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2021-11-29 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2022-06-28 (Actual)

PRIMARY OUTCOMES:
Mean change in maximal voluntary isometric force of the knee extensors from pre-intervention up to 72 hours post-intervention | Immediately pre-intervention, immediately post-intervention, 24 hours post-intervention, 48 hours post-intervention, 72 hours post-intervention
  The change in the maximum amount of voluntary isometric force produced by the knee extensors, assessed via a series of maximal voluntary contractions performed at 90 degrees of knee flexion (extension = 0 degrees).

SECONDARY OUTCOMES:
Mean change in the joint angle-torque curve of the knee extensors from pre-intervention up to 72 hours post-intervention | Immediately pre-intervention, immediately post-intervention, 24 hours post-intervention, 48 hours post-intervention, 72 hours post-intervention
  The change in the joint angle-torque curve of the knee extensors, assessed using a series of maximal isokinetic contractions performed from 90 to 0 degrees of knee flexion at an angular velocity of 45 degrees per second.
Mean change in plasma creatine kinase from pre-intervention up to 72 hours post-intervention | Immediately pre-intervention, 24 hours post-intervention, 48 hours post-intervention, 72 hours post-intervention
  The change in plasma creatine kinase assessed via a commercially-available assay kit.
Mean change in pain-free range of motion of the knee extensors from pre-intervention up to 72 hours post-intervention | Immediately pre-intervention, 24 hours post-intervention, 48 hours post-intervention, 72 hours post-intervention
  "Pain-free range of motion of the knee extensors" describes the degree of passive knee flexion the participant can achieve until they reach a point of self-perceived soreness. The assessment involves the investigator progressively moving the shank of the participant into further knee flexion until the participant experiences noticeable discomfort, at which the knee joint angle will be measured using a goniometer.
Mean change in muscle thickness of the rectus femoris and vastus lateralis from pre-intervention up to 72 hours post-intervention | Immediately pre-intervention, 24 hours post-intervention, 48 hours post-intervention, 72 hours post-intervention
  The change in muscle thickness of the rectus femoris and vastus lateralis when measured using B-mode ultrasound at 50 percent total femur length. Muscle thickness will be defined as the mean perpendicular distance between the deep and superficial aponeuroses at the proximal, central, and distal portions of the acquired images.
Mean change in perceived muscle soreness from pre-intervention up to 72 hours post-intervention | Immediately pre-intervention, 24 hours post-intervention, 48 hours post-intervention, 72 hours post-intervention
  The change in perceived lower-body muscle soreness when assessed at rest and during voluntary flexion and extension of the knee. Soreness at rest and during motion will be quantified separately using a 100 mm visual analogue scale titled "Visual Analogue Scale for Muscle Soreness". Participants will be asked to mark their perceived soreness at any point along a horizonal line ranging from 0 mm (no soreness at all) to 100 mm (most soreness ever experienced). Scores will be rounded to the nearest 1 mm.

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Gapper, Principal Investigator — University of Surrey
Locations (1):
- University of Surrey, Guildford, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Data spreadsheet will be available upon request from the principle investigator.

REFERENCES:
- [Background] Patterson SD, Hughes L, Warmington S, Burr J, Scott BR, Owens J, Abe T, Nielsen JL, Libardi CA, Laurentino G, Neto GR, Brandner C, Martin-Hernandez J, Loenneke J. Blood Flow Restriction Exercise: Considerations of Methodology, Application, and Safety. Front Physiol. 2019 May 15;10:533. doi: 10.3389/fphys.2019.00533. eCollection 2019. PMID 31156448
- [Background] Lixandrao ME, Ugrinowitsch C, Berton R, Vechin FC, Conceicao MS, Damas F, Libardi CA, Roschel H. Magnitude of Muscle Strength and Mass Adaptations Between High-Load Resistance Training Versus Low-Load Resistance Training Associated with Blood-Flow Restriction: A Systematic Review and Meta-Analysis. Sports Med. 2018 Feb;48(2):361-378. doi: 10.1007/s40279-017-0795-y. PMID 29043659
- [Background] de Queiros VS, Dos Santos IK, Almeida-Neto PF, Dantas M, de Franca IM, Vieira WHB, Neto GR, Dantas PMS, Cabral BGAT. Effect of resistance training with blood flow restriction on muscle damage markers in adults: A systematic review. PLoS One. 2021 Jun 18;16(6):e0253521. doi: 10.1371/journal.pone.0253521. eCollection 2021. PMID 34143837
- [Background] Hyldahl RD, Hubal MJ. Lengthening our perspective: morphological, cellular, and molecular responses to eccentric exercise. Muscle Nerve. 2014 Feb;49(2):155-70. doi: 10.1002/mus.24077. Epub 2013 Dec 3. PMID 24030935